CLINICAL TRIAL: NCT01527851
Title: Impact of Excess Skin on the Practice of Physical Activity in Women Who Underwent Bariatric Surgery and Exploration of the Benefits of Plastic Surgery
Brief Title: Excess Skin and Physical Activity
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-France Langlois, Principal investigator, Université de Sherbrooke
Other Study IDs: 11-190
Record Dates: First submitted 2012-02-01; First posted 2012-02-07 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Post-bariatric surgery; Excess skin; Physical fitness; Physical activity; Barriers to physical activity; Plastic surgery; Quality of life; Self-esteem
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction: Currently, bariatric surgery appears to be the most effective treatment to improve the health of morbidly obese population. However, the massive weight loss induced by this intervention can create excess loose skin in various parts of the body contributing to the feeling of failure in their desire to feel better in some patients. Several studies show that people are once again disappointed and dissatisfied with their body appearance due to the mass of unsightly loose skin that disrupts their quality of life. However, very few studies have focused on the barriers that this excess skin could create in everyday physical activity. The aim of the investigators pilot study is to assess the impact of excess skin on the practice of physical activity in women who underwent bariatric surgery and evaluate if there is a relationship between physical activity and the level and location of excess skin. Also, the investigators will explore, the benefits of plastic surgery in patients who had this intervention.

Materials and methods: About twenty women who underwent bariatric surgery and a dozen who had subsequent plastic surgery will be included in this pilot study. Anthropometry, weight loss post bariatric and plastic surgery, motivational stage on the practice of physical activity, usual practice of physical activity, functional and physical ability, perceived benefits and barriers of physical activity, self-esteem and quality of life will be assessed. After analyzing the results, a group discussion will be established to further evaluate the impact of excess skin on the practice of physical activity. The evaluation will be identical for monitoring the effects of plastic surgery but the discussion group will also address the benefits and satisfaction related to plastic surgery.

Expected results: Excess skin could be a barrier to physical activity by limiting the functional and physical capacity. Thus, plastic surgery could improve the practice of physical activity with a direct improvement of functional discomfort, the subjects' motivation to be physically active, perceived benefits and barriers to physical activity, self-esteem and quality of life.

Issue project: This pilot project will generate data that will allow us, depending on the relevance of the results, to continue the investigators investigation with a larger cohort.

ELIGIBILITY:
Inclusion Criteria:

* have underwent bariatric surgery more than 1 year ago
* had a weight loss of at least 20% after bariatric surgery
* had a weight change of less than 5 kg in the last 3 months
* woman > 18 years old
* have read and given consent

Inclusion Criteria for the group post-plastic:

* have underwent a plastic surgery at least 6 months ago

Exclusion Criteria:

* medical contraindication for physical activity
* major functional limitations : failure to realize different tests
* intellectual disability and/or neuropsychological disease
* not being able to speak or understand french

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of 20 people who underwent bariatric surgery and a group of 10 people who underwent bariatric surgery and one or several plastic surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10-21 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Physical activity pratice | Initial
  Inconvenience during physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Baillot A, Asselin M, Comeau E, Meziat-Burdin A, Langlois MF. Impact of excess skin from massive weight loss on the practice of physical activity in women. Obes Surg. 2013 Nov;23(11):1826-34. doi: 10.1007/s11695-013-0932-0. PMID 23620304